CLINICAL TRIAL: NCT07393256
Title: Probiotic and Synbiotic Supplementation for Constipation-related Outcomes in Children With Cerebral Palsy: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Probiotics on Constipation and Weight in CP
Acronym: cerebral palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Aybegum Kalyoncu Aycenk, Assistant Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/82
Record Dates: First submitted 2026-01-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Constipation; Probiotic
Keywords: cerebral palsy; constipation; children; probiotics; Lactobacillus reuteri; Lactobacillus rhamnosus; inulin
MeSH Terms: conditions — Cerebral Palsy; Constipation | interventions — Prebiotics; Inulin

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, double-blind, randomized controlled trial with three parallel groups. Participants with cerebral palsy and chronic constipation are randomly assigned in equal numbers to one of three groups: (1) Lactobacillus reuteri, (2) Lactobacillus rhamnosus supplemented with prebiotic inulin, or (3) control. Each participant receives only one intervention throughout the 28-day study period. Neither the participants, caregivers, nor the investigators responsible for assessment are aware of group allocation.
Who Masked: Participant, Investigator
Masking Description: Both participants (caregivers and children) and the investigators responsible for data collection and outcome assessment were blinded to group assignments. The probiotic products and packaging were identical in appearance, taste, and labeling. The randomization code was held by an independent coordinator and was not revealed to the study team until data analysis was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lactobacillus reuteri group (Experimental): Participants receive Lactobacillus reuteri supplement daily for 28 days.
  Interventions: Dietary Supplement: Lactobacillus Reuteri Oral Solution [BioGaia]
- Lactobacillus rhamnosus + Prebiotic (Inulin) group (Experimental): Participants receive Lactobacillus rhamnosus with prebiotic inulin daily for 28 days.
  Interventions: Dietary Supplement: Lactobacillus Rhamnosus; Dietary Supplement: Prebiotic (inulin)
- Control group (No Intervention): Participants receive standard dietary management (no probiotic supplementation).

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri Oral Solution [BioGaia] — Participants receive *Lactobacillus reuteri* supplement once daily for 28 days.
  Arms: Lactobacillus reuteri group
Dietary Supplement: Lactobacillus Rhamnosus — Lactobacillus rhamnosus is administered as part of a single synbiotic product that also contains the prebiotic inulin. The synbiotic formulation is provided as one commercially available product and is administered once daily for 28 days.
  Arms: Lactobacillus rhamnosus + Prebiotic (Inulin) group
Dietary Supplement: Prebiotic (inulin) — Inulin is administered as part of the same single synbiotic product that contains Lactobacillus rhamnosus. The synbiotic formulation is provided as one commercially available product and is administered once daily for 28 days.
  Arms: Lactobacillus rhamnosus + Prebiotic (Inulin) group

SUMMARY:
The goal of this clinical trial is to learn whether using Lactobacillus reuteri or a prebiotic-containing Lactobacillus rhamnosus supplement helps to improve constipation and weight gain in children with cerebral palsy (CP). It will also examine the safety and tolerability of these probiotic products.

The main questions it aims to answer are:

Do these probiotic supplements improve bowel movement frequency and stool consistency?

Do they support better weight gain and nutritional status in children with CP?

Are there any side effects or tolerability issues during treatment?

Researchers will compare Lactobacillus reuteri with prebiotic-enriched Lactobacillus rhamnosus in a randomized, double-blind, controlled design.

Participants will:

Take one of the probiotic products daily for 28 days

Visit the clinic at the beginning and end of the study for measurements and stool testing

Have their caregivers keep a stool diary using the Bristol stool scale

DETAILED DESCRIPTION:
ClinicalTrials.gov Study Record Example Title The Effect of Using Lactobacillus reuteri and Prebiotic-Containing Lactobacillus rhamnosus Strains on Constipation and Weight Gain in Children with Cerebral Palsy: A Prospective Randomized Controlled Study ________________________________________ Brief Summary This clinical trial aims to determine whether daily supplementation with Lactobacillus reuteri or a prebiotic-enriched Lactobacillus rhamnosus formula can improve constipation and weight gain in children with cerebral palsy (CP). Constipation is a common problem in children with CP due to impaired intestinal motility and disruption of the gut microbiota. The study will compare the effects and safety of two probiotic products over a 28-day period.

________________________________________ Detailed Description Cerebral palsy (CP) is a non-progressive neurodevelopmental disorder characterized by impairments in movement and posture. Gastrointestinal complications, particularly chronic constipation and inadequate weight gain, are frequently observed in this population and may significantly affect quality of life. Altered intestinal motility, limited physical activity, and gut microbiota dysbiosis are considered key contributors to bowel dysfunction in children with CP.

Probiotics have been proposed as a supportive therapeutic approach for gastrointestinal symptoms through modulation of intestinal microbiota, enhancement of barrier function, and regulation of bowel motility. Lactobacillus reuteri and Lactobacillus rhamnosus are among the most commonly studied probiotic strains with documented benefits in pediatric gastrointestinal disorders. The addition of prebiotics such as inulin may further enhance probiotic efficacy by promoting the growth of beneficial bacteria.

This prospective, randomized, double-blind, controlled study is designed to evaluate the effects of daily probiotic supplementation on bowel habits and growth parameters in children with cerebral palsy. Eligible participants are allocated to one of three parallel intervention arms and followed for a 28-day treatment period.

Clinical assessments are conducted at baseline and at the end of the intervention period. Anthropometric measurements are obtained using standardized techniques. Stool samples are collected for laboratory analysis, and stool consistency is evaluated using a validated scoring system. Caregivers maintain a daily stool diary to document bowel movement frequency and gastrointestinal symptoms throughout the study period.

The study evaluates changes in bowel function and growth-related parameters over time, as well as the safety and tolerability of the probiotic formulations. Adverse events and treatment adherence are monitored throughout follow-up. This study aims to provide evidence on whether probiotic supplementation represents a safe and effective supportive strategy for managing constipation and improving nutritional outcomes in children with cerebral palsy.

________________________________________ Study Type Interventional (Clinical Trial) Study Design

* Allocation: Randomized
* Intervention Model: Parallel Assignment
* Masking: Double-blind (Participant, Investigator)
* Primary Purpose: Treatment ________________________________________ Estimated Enrollment (Insert total number, e.g., n = 90 participants)

Official Title The Effect of Using Lactobacillus reuteri and Prebiotic-Containing Lactobacillus rhamnosus Strains on Constipation and Weight Gain in Children with Cerebral Palsy: A Prospective Randomized Controlled Study ________________________________________ Arms and Interventions Arm 1: Lactobacillus reuteri Participants receive Lactobacillus reuteri daily for 28 days. Arm 2: Lactobacillus rhamnosus + Prebiotic (Inulin) Participants receive a probiotic containing Lactobacillus rhamnosus with prebiotic inulin daily for 28 days.

Arm 3: Control Group Participants receive standard dietary management for constipation.

________________________________________ Primary Outcome Measures

1. Change in defecation frequency [Time Frame: Baseline and Day 28]
2. Change in stool consistency (Bristol Stool Scale) [Time Frame: Baseline and Day 28] ________________________________________ Secondary Outcome Measures

<!-- -->

1. Change in body weight and BMI [Time Frame: Baseline and Day 28]
2. Stool pH level [Time Frame: Baseline and Day 28]
3. Caregiver-reported gastrointestinal symptoms [Time Frame: Throughout 28-day follow-up]
4. Incidence of adverse events [Time Frame: Throughout 28-day follow-up]

   ________________________________________ Eligibility Criteria

   Inclusion Criteria:
   * Children aged 2-18 years
   * Diagnosed with cerebral palsy (GMFCS levels III-V)
   * Chronic constipation meeting Rome IV criteria
   * Stable medical condition and able to take oral or enteral feeding

   Exclusion Criteria:

   • Degenerative neurological diseases
   * Congenital gastrointestinal malformations
   * Inflammatory bowel disease or metabolic disorders
   * Kidney failure
   * Antibiotic, probiotic, or prebiotic use within one month before enrollment
   * Poor adherence (<95%) or hospitalization during study period ________________________________________ Study Start Date January 2023 Estimated Study Completion Date February 2025 ________________________________________ Location Ordu University Faculty of Medicine, Departments of Pediatric Surgery, Pediatrics, and Pediatric Neurology, Ordu University Training and Research Hospital, Ordu, Turkey

   Sponsors and Collaborators

   • Sponsor: Ordu University Faculty of Medicine, Department of Pediatric Surgery

   • Collaborators: Department of Pediatrics and Division of Pediatric Neurology

   • Product Support: Nestlé (Inulin-Enriched Lactobacillus rhamnosus formulation)

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 18 years
* Clinical diagnosis of cerebral palsy
* Gross Motor Function Classification System (GMFCS) levels III, IV, or V
* Chronic constipation diagnosed according to Rome IV criteria
* Stable medical condition
* Ability to receive oral or enteral nutrition

Exclusion Criteria:

* Cerebral palsy due to degenerative neurological disorders
* Constipation due to a known organic cause
* Congenital gastrointestinal tract malformations
* Inflammatory bowel disease
* Metabolic diseases
* History of kidney failure
* Use of antibiotics, probiotics, or prebiotics within one month prior to enrollment
* Anticipated poor adherence to the study protocol
* Requirement for hospitalization during the study period

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Change in stool consistency (Bristol Stool Scale) | Baseline and Day 28
  Stool form assessed using the Bristol Stool Scale (types 1-7). Higher scores reflect softer stool consistency.
Change in defecation frequency | Baseline and Day 28
  Number of bowel movements per week, recorded in caregiver stool diaries. Increase in defecation frequency indicates improvement in constipation.
Change in Stool Consistency (Bristol Stool Scale) | Baseline and Day 28
  Change in stool consistency assessed using the Bristol Stool Scale (types 1-7). Improvement is defined as an increase in Bristol Stool Scale score from baseline to Day 28.

SECONDARY OUTCOMES:
Change in stool pH | Baseline and Day 28
  Stool samples analyzed for pH using a standard test kit to evaluate intestinal microbiota activity.
Change in body weight | Baseline and Day 28
  Change in body weight measured in kilograms. An increase indicates improved nutritional status.
Change in body mass index (BMI) | Baseline and Day 28
  Change in body mass index calculated as weight in kilograms divided by height in meters squared (kg/m²).
Change in mid-arm circumference | Baseline and Day 28
  Change in mid-arm circumference measured in centimeters as an indicator of muscle mass and nutritional status.
Change in heel-to-knee length | Baseline and Day 28
  Change in heel-to-knee length measured in centimeters as an indicator of linear growth.
Caregiver-reported gastrointestinal symptoms | Throughout 28-day follow-up
  Caregiver-reported presence and frequency of gastrointestinal symptoms, including gagging, vomiting, retching, bloating, and feeding intolerance, recorded using a daily symptom diary. No composite symptom score is calculated.
Incidence of adverse events | Throughout 28-day follow-up
  Number and type of any adverse or unexpected reactions observed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Aybegum Kalyoncu Aycenk, Assistant Professor, Study Director — ORDU UNIVERSITY, FACULTY OF MEDICINE, DEPARTMENT OF PEDIATRIC SURGERY
Locations (1):
- Ordu University Faculty of Medicine, Department Of Pediatric Surgery, Ordu, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share individual participant data outside of the research team due to ethical considerations and patient confidentiality.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT07393256/Prot_ICF_000.pdf